CLINICAL TRIAL: NCT05242081
Title: Efficacy and Safety of Opioid-free Anesthesia With Propofol Combined With S-ketamine in Laparoscopic Cholecystectomy: a Multicenter, Randomized, Controlled, Non-inferiority Clinical Study (SKOF - LC)
Brief Title: Study on Opioid-free Anesthesia Protocol With S-ketamine and Propofol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-SR-480
Record Dates: First submitted 2022-01-13; First posted 2022-02-16 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Opioid Use, Unspecified; S-ketamine
MeSH Terms: interventions — Esketamine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-ketamine (Experimental)
  Interventions: Drug: S-ketamine
- Sufentanil (Active Comparator)
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: S-ketamine — S-ketamine 0.5mg/kg for induction and 0.2mg/kg/h for maintenance
  Arms: S-ketamine
Drug: Sufentanil — Sufentanil 0.2-0.3μg/kg for induction and remifentanil 0.05-0.15μg/kg/min for maintenance
  Arms: Sufentanil

SUMMARY:
The purpose of this study was to observe the effects of opioid-free anesthesia with S-ketamine on postoperative analgesia and perioperative hemodynamics in short surgical operations, and to explore the effects of S-ketamine on postoperative awakening time and extubation time, nausea and vomiting, hypoxemia, and delirium.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 18 years to 65 years
2. American society of anesthesiologists physical status classification I-II
3. Patients scheduled for elective laparoscopic cholecystectomy
4. Willing to sign informed consent

Exclusion Criteria:

1. Allergic to narcotic drugs;
2. Surgical history within the past 1 month;
3. patients with neurological diseases or mental disorders;
4. Unable to understand numerical rating Scale (NRS);
5. patients with untreated or poorly controlled hypertension (arterial hypertension, resting systolic/diastolic blood pressure over 180/100mmHg);
6. patients with untreated or undertreated hyperthyroidism;
7. Patients with unstable angina pectoris or myocardial infarction in the past 6 months;
8. When intraocular pressure is high (glaucoma) and penetrating ocular trauma, intraocular pressure cannot rise.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 980 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The probability of numerical rating scale (NRS) score being less than or equal to 3 when leaving the Postanesthesia Care Unit (PACU) | 1 day of the surgery
  The probability of numerical rating scale (NRS) score being less than or equal to 3 when leaving the Postanesthesia Care Unit (PACU)

SECONDARY OUTCOMES:
The area under the curve (AUC) of mean arterial pressure (MAP) within 10 minutes after induction is lower than the baseline mean arterial pressure (MAP 3 minutes before induction). | From the date of the beginning of anesthesia until the date of the end of anesthesia, assessed up to 2 days
  The area under the curve (AUC) of mean arterial pressure (MAP) within 10 minutes after induction is lower than the baseline mean arterial pressure (MAP 3 minutes before induction).
herat rate and blood pressure during the surgery every 5 minutes | From the date of the beginning of anesthesia until the date of the end of anesthesia, assessed up to 2 days
Total dosage of anesthesia drug | From the date of the beginning of anesthesia until the date of the end of anesthesia, assessed up to 2 days
Total dosage of vasoactive agents | From the date of the beginning of anesthesia until the date of the end of anesthesia, assessed up to 2 days
The duration of surgery | From the date of the beginning of surgery until the date of the end of surgery, assessed up to 2 days
Time until awake | From the end of anesthesia until awake, assessed up to 2 days
Time to removal of tracheal intubation | From the end of anesthesia until the time of removal of tracheal intubation, assessed up to 2 days
Incidence of postoperative nausea and vomiting | 48 hours after the surgery
Incidence of postoperative delirium | 48 hours after the surgery
Incidence of hypoxemia | 48 hours after the surgery
Postoperative first analgesia demand | From the end of anesthesia until the date of first demand of analgesia drugs, assessed up to 1 week
  The first time that the patient ask for analgesia
numerical rating scale (NRS) pain score | 24 hours and 48 hours after the surgery
Postoperative hospital stay | From the date of the surgery until the date being discharged from hospital, up to 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China